CLINICAL TRIAL: NCT02391844
Title: Open-Label Parallel Group Flexible Dosing & Titration Study to Evaluate the Efficacy, Safety of Oxycodone/APAP Extended Release Formulation Xartemisxr® in the Management of Post-Operative Pain Following Outpatient Arthroscopic Knee Surgery
Brief Title: Open-Label Study of Oxycodone/APAP to Treat Post-Operative Pain Following Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Clinical Research Institute (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK795-ICRI-001
Record Dates: First submitted 2014-05-15; First posted 2015-03-18 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-11

CONDITIONS: Disorder of Knee
Keywords: Knee; Post-Operative Pain; Xartemis
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone (Other): Xartemis XR - Oxycodone with Acetaminophen Extended Release Tablet
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Oxycodone with Acetaminophen Extended Release
  Other Names: Xartemix XR

SUMMARY:
This is a pilot trial using this product in patients for the management of pain after outpatient arthroscopic knee surgery. This is an open-label study and the two active ingredients are well known pharmacologic entities.

DETAILED DESCRIPTION:
The objective of this single center is to evaluate the safety and efficacy of Oxycodone Extended Release (MNK-795) in postoperative pain following common musculoskeletal surgical procedures. Knee surgery being the most common surgery performed in the US, the investigators chose the model. The investigators also want to look at the flexible-dosing and titration which is the common way pain managed by clinicians. This is an open-label study of MNK 795 to be described in the procedures section.

Primary endpoint:

• Change in pain from baseline (before taking the first dose of study medication) measured on NRS

Secondary endpoints:

* Patient/Investigator Global assessment of treatment satisfaction
* Safety evaluation with adverse event monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-75 who underwent an orthopedic outpatient surgical procedure of their knee
2. Read and understand English and comprehend the procedures associated with participating in a clinical trial.
3. Signed an IRB approved consent form and HIPAA authorization
4. Patients with a pain intensity score of 4 or above on the 0-10 numerical rating scale (0 is no pain, 10 is the worst pain imaginable)

Exclusion Criteria:

1. Participants in any other clinical trial in the last 30 days or currently enrolled in a clinical trial
2. Allergy to Oxycodone or Acetaminophen.
3. Uncontrolled pain or other pain conditions that may interfere with evaluation
4. Pregnant women
5. Women who are trying to become pregnant
6. Women who are breastfeeding
7. Patient who is deemed to be medically unstable by the principal investigator
8. History of Alcohol, opioid or substance abuse in the last 2 yrs
9. History of sleep apnea that requires CPAP
10. History of serious respiratory illness
11. History of Gastric bypass
12. Prior use of opiates at doses higher than 90mg Morphine equivalent dosing
13. Will limit the study medication to 4 tab at each dosing and to total dose of 8 tab for 24 hrs. Subjects needing doses higher than that, based on their current opioid dose, will not be enrolled or discontinued

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in pain Scores on the Numerical Rating Scale | Baseline to Week 4
  Change in pain Scores on the Numerical Rating Scale from baseline (before taking the first dose of study medication) through 4 week study participation.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Screening to Week 4
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

OTHER OUTCOMES:
Assessment of Treatment Satisfaction | 1 Week, 2 Weeks, and 4 Weeks Post Dose
  Patient/Investigator Global assessment of treatment satisfaction will be completed 3 follow-up visits after screening.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute
Locations (1):
- International Clinical Research Institute, Overland Park, Kansas, United States